CLINICAL TRIAL: NCT02808442
Title: A Phase 1, Open Label, Non-comparative Study to Evaluate the Safety and the Ability of UCART19 to Induce Molecular Remission in Paediatric Patients With Relapsed/Refractory B-cell Acute Lymphoblastic Leukaemia
Brief Title: Study of UCART19 in Pediatric Patients With Relapsed/Refractory B Acute Lymphoblastic Leukemia
Acronym: PALL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCART19_02 (CL1-68587-001); 2015-004293-15 (EudraCT Number)
Record Dates: First submitted 2016-06-16; First posted 2016-06-21 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Refractory B-cell Acute Lymphoblastic Leukemia; Relapsed B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- UCART19 (Experimental)
  Interventions: Biological: UCART19

INTERVENTIONS:
Biological: UCART19
  Other Names: S68587

SUMMARY:
This study aims to evaluate the safety and feasibility of UCART19 to induce molecular remission in pediatric patients with relapsed or refractory CD19-positive B-cell acute lymphoblastic leukemia (B-ALL).

ELIGIBILITY:
Inclusion Criteria:

* Patient with relapsed or refractory CD19-positive B-acute lymphoblastic leukaemia (B-ALL) who have exhausted alternative treatment options.
* Estimated life expectancy ≥ 12 weeks
* Lansky (age < 16 years at the time of assent/consent) or Karnofsky (age ≥ 16 years at time of assent/consent) performance status ≥ 50

Exclusion Criteria:

* Burkitt leukemia
* CD19-negative B-cell leukemia
* Active Central Nervous System (CNS) leukemia
* Active acute or chronic Graft-versus-Host Disease (GvHD) requiring systemic use therapy within 4 weeks before UCART19 infusion
* Patients with autoimmune disease requiring systemic immunosuppression therapy that cannot be stopped
* History of CRS grade 4 related to previous CAR T cell therapy
* Contraindication to Alemtuzumab administration

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2020-09-17 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events | From inclusion to Month 12
  Adverse events assessed according to NCI-CTCAE v5.0 criteria

SECONDARY OUTCOMES:
Molecular Remission Rate | At Day 28 after the first UCART19 infusion
  Proportion of patients in whom a molecular Complete Remission (CR) or a Complete Remission with incomplete blood recovery (CRi) is observed (i.e. a CR or CRi combined to a Minimal residual disease <10-4).

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Hôpital Robert-Debré, Paris, France
- Hospital San Juan De Dios, Barcelona, Spain
- UCL Great Ormond Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- [Result] Benjamin R, Graham C, Yallop D, Jozwik A, Mirci-Danicar OC, Lucchini G, Pinner D, Jain N, Kantarjian H, Boissel N, Maus MV, Frigault MJ, Baruchel A, Mohty M, Gianella-Borradori A, Binlich F, Balandraud S, Vitry F, Thomas E, Philippe A, Fouliard S, Dupouy S, Marchiq I, Almena-Carrasco M, Ferry N, Arnould S, Konto C, Veys P, Qasim W; UCART19 Group. Genome-edited, donor-derived allogeneic anti-CD19 chimeric antigen receptor T cells in paediatric and adult B-cell acute lymphoblastic leukaemia: results of two phase 1 studies. Lancet. 2020 Dec 12;396(10266):1885-1894. doi: 10.1016/S0140-6736(20)32334-5. PMID 33308471
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: Study-level clinical trial data — https://clinicaltrials.servier.com/